CLINICAL TRIAL: NCT06769074
Title: Assessment of Role of Platelet Rich Plasma in Managing Women with Mixed Urinary Incontinence
Brief Title: Assessment of Platelet Rich Plasma Injection in Managing Female Patients Complaining of Mixed Urinary Incontinence (PRP)
Acronym: PRP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 782/29-oct-2024
Record Dates: First submitted 2024-12-29; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Mixed Urinary Incontinence
Keywords: Mixed urinary incontinence; Platelet rich plasma; stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PRP injection at midurethra with PRP instillation into urinary bladder (Experimental): A-PRP was injected into the anterior vaginal mucosa around the mid-urethral area, which was approximately 1 cm below the urethral meatus and had a depth of about 1.5 cm; 2 mL were injected underneath the mid-urethral area and 1.5 mL was injected on either side of the urethra
  *10ml PRP used to instill intravesical for urgency urinary incontinence by urethral catheter
  Interventions: Biological: Platelet Rich Plasma

INTERVENTIONS:
Biological: Platelet Rich Plasma — PRP injection into the midurethra and its instillation into urinary bladder

SUMMARY:
The goal of this clinical trial is to assess the efficacy of platelet-rich plasma (PRP) for the treatment of mixed urinary incontinence determine .The main question it aims to answer whether PRP is it safe and effective in managing mixed urinary incontinence? Researchers will assess efficacy of PRP in both stress and urgency incontinence treatment

Participants will:

* Undergo PRP injection in to mid urethra , and installation into bladder every 1 month for 3 month
* Visit the clinic once every 1 month for checkups and urodynamic study after 3 month, and 4 month after last installation

DETAILED DESCRIPTION:
All patients will be subjected to:

* An informed consent will be taken from every patient.
* Complete history taking:

  * Personal history
  * Any complaint.
  * Past medical and past surgical history.
  * Family history.
  * Severity of incontinence by International consultation on incontinence questionnaire- short form (ICIQ-SF), OAB symptom score ,Cough stress test

    *Complete physical examination.
  * General examination: Vital signs (Blood pressure, Temperature, Heart rate, Respiratory rate).
  * neurological examination: gait, perineal sensation, bulbocavernous reflex, cognitive status
  * abdominal examination : distended bladder, masses , hernia, DRE
  * Pelvic examination: vaginal atrophy, skin excoriation, vault examination, organ prolapse, pelvic floor muscle strength , cough test, Q tip test, Marshall test
  * urodynamics done for documentation of detrusor overactivity before and after PRP installation after 3rd instillation and 4 m after last instillation

    * patient is placed in the dorsal lithotomy position
    * PRP is obtained from a sample of patients' blood drawn at the time of treatment
    * A 30 cc venous blood draw will yield 3-5 cc of PRP
    * The blood draw occurs with the addition of an anticoagulant, such as citrate dextrose A( .5 ml)to prevent platelet activation prior to its use
    * in room temp 21-24 to avoid activation of platelet
    * a specialized 'table top cold centrifuge' device to centrifugate the sample
    * After centrifugation, each vial was confirmed to contain three layers from top to bottom, namely, the platelet pellet, gel, and red blood cells. The platelet pellet was remixed with the supernatant by inverting the tubes gently 5-10 times.
    * A-PRP was injected into the anterior vaginal mucosa around the mid-urethral area, which was approximately 1 cm below the urethral meatus and had a depth of about 1.5 cm; 2 mL were injected underneath the mid-urethral area and 1.5 mL was injected on either side of the urethra
    * 10ml PRP used to instill intravesical for urgency urinary incontinence by urethral catheter
    * patient received four injections of PRP at monthly intervals
    * follow up done after 3rd instillation and 4 months after finishing injections
    * follow up done by subjective symptoms as previous scoring system and objective by Urodynamics

ELIGIBILITY:
Inclusion Criteria:

* Women with MUI ( mild and moderate degree of stress incontinence)
* Age between 20 to 60 years -

Exclusion Criteria:

* intrinsic sphincteric deficiency (ISD)
* Pregnancy
* Sepsis
* Acute and chronic infections
* Chronic liver disease
* Anti-coagulation therapy
* History of malignancy
* Under anti-platelet agent treatment

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-28 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of females with treatment-related improvement of mixed urinary incontinence after receiving platelet-rich plasma (PRP) injection and instillation. | From enrollment to the end of intervention at 6 month "
  Treatment -related improvement of urinary incontinence is assessed using:
  * International consultation on incontinence questionnaire- short form (ICIQ-SF).
  * OAB symptom score.
  * Cough stress test.
  * Urodynamics.
    1. ICIQ-Sf questionnaire before and after treatment: Scoring scale: 0-21, minimum 0, maximum 21. A higher score indicates greater impairment from incontinence.
    2. OAB symptom score: has a maximum score of 15 with more weight assigned to urgency and urgency incontinence than on frequency. Higher score indicates greater impairment from incontinence.
    3. Urodynamics: for assessment of of detrusor over-activity before and after treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Zagazig University, Egypt
  - Zagazig university hospital , Egypt, Zagazig